CLINICAL TRIAL: NCT01880918
Title: Multi Center, Observational, Retrospective Data Collection of Patients Treated With the ColonRing in Routine Clinical Practice. This Study to Continue RETROPRESS Study ID NCT01301417
Brief Title: A RETROspective Data Collection of comPRESSion Anastomosis Using the ColonRing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: novoGI (Industry)
Responsible Party: Sponsor
Other Study IDs: RETROPRESS, CLPR-43-11-01
Record Dates: First submitted 2013-06-16; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Diverticulum, Colon; Colorectal Neoplasms; Crohn Disease; Colitis, Ulcerative; Colostomy; Ileostomy - Stoma; Rectal Prolapse; Intestinal Polyposis; Lymphoma; Endometriosis; Intestinal Volvulus
Keywords: Compression Anastomosis
MeSH Terms: conditions — Diverticulum, Colon; Colorectal Neoplasms; Crohn Disease; Colitis, Ulcerative; Rectal Prolapse; Intestinal Polyposis; Lymphoma; Endometriosis; Intestinal Volvulus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ColonRing: The ColonRing device is intended to be used for the creation of intestinal anastomoses in colorectal surgery in both open and laparoscopic surgeries. This indication is within the currently cleared indication of the ColonRing device, which has been cleared by the US FDA and carries the CE Mark for use throughout the alimentary trct for the creation of circular end-to-end, side-to-end or side-to-side anastomosis.

SUMMARY:
The proposed study is a post marketing, observational, retrospective data collection intended to gather and record data on patients treated with the ColonRing device in routine clinical practice at 4-6 centers. The data will assist in future evaluating the performance of the ColonRing device in regards to the creation of a colorectal anastomosis in Low Anterior Resection procedures.

Hypothesis: The performance of the ColonRing, determined by the rate of complications, will be within the acceptable range reported in the literature for alternative treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was > 18 years old at time of procedure
2. Patient underwent a technically successful open or laparoscopic colorectal, Low Anterior Resection procedure with the creation of an anastomosis using the ColonRing™
3. Patient treated in routine clinical practice
4. Patient underwent his/her first follow-up visit within two months post-surgery

Exclusion Criteria:

No exclusion criteria have been defined for this data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent a laparoscopic or open Low Anterior resection with the creation of an anastomosis using the ColonRing in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The rate of anastomotic leakage. | 6 weeks after the procedure
  Anastomotic leakage is defined as evidence of a defect in the intestinal wall integrity at the anastomotic site leading to a communication between the intra and extra luminal compartments.

SECONDARY OUTCOMES:
Rate of other device related complications and measures during hospitalization and post procedure. | 6 weeks after the procedure.
  The Following complications will be examined:
  Bleeding. Stricture (either clinical evidence of a stricture or the inability to pass a 12 mm sigmoidoscope through the anastomosis in a procedure that does not include a diversion). Septic complication (including wound infection, pelvic infection, peritonitis, abscess) Readmission, re-operation, death within two months of the procedure Extra colonic complications (including urinary infection, urinary retention, DVT, pneumonitis, pulmonary embolism, cardiac, injury to other organs - e.g. spleen, ureter)
  The following post operative measures will be reported:
  Hospitalization duration (two dates will be recorded: ready for discharge and discharge). The latter noting where the patient was discharged to - e.g. nursing home or home. First day to first postoperative flatus. First day to first postoperative bowel movements. First day of first postoperative toleration of liquids and solids (time to "keeping them down")

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Florida Hospital, Center for Colon & Rectal Surgery, Atlamonte Springs, Florida
  - 18308 Murdock Circle, Suite 108, Port Charlotte, Florida
  - CoxHealth Hospital, Colorectal Department, Springfield, Missouri